CLINICAL TRIAL: NCT06155630
Title: 3D Printing vs Traditional Workflow for the Fabrication of Mandibular Implant Overdentures: A Randomized Cross-over Clinical Trial
Brief Title: 3D Printing for the Fabrication of Mandibular Implant Overdentures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1680-2022; 1744-2023 (Other Grant/Funding Number: ITI)
Record Dates: First submitted 2023-11-22; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Edentulous Mouth; Edentulous Jaw
Keywords: 3D printing; Implant overdenture; clinical trial
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printed mandibular implant overdenture (Experimental): First appointment: The first visit will consist of scanning the patients' existing upper complete denture and lower mandibular implant overdenture by using a desktop scanner. In the lab, the .stl files will be 3D printed using a DLP 3D printer. Second clinical appointment: the interim printed dentures will be adjusted with wax for the desired lip support and VD. Secondary impressions will be taken to refine fit. Maxillary and mandibular interim printed dentures will be scanned separately and together with an intraoral scanner. Patient's face will also be scanned by a face scanner. 2nd lab session: .stl files will be superimposed for the digital pathway. Teeth and denture bases will be designed virtually. Dentures bases will be manufactured by a DLP 3D printer with Dentca Resin. Dentures will receive Dentsply Portrait 3D teeth. Dentures will be finished and polished, and sandblasted in the attachment sockets. 4th appointment: denture delivery.
  Interventions: Other: mandibular implant-overdenture
- traditional mandibular implant overdenture (Active Comparator): The first visit will be the same. For the conventional pathway, the 2nd lab session will consist of pouring the impressions (type 4 stone), mounting the casts in arcon semi-adjustable articulator, removing the printed teeth, and replacing it with wax rim and acrylic tooth setup (Dentsply Portrait - same shape, size and shade used for 3D printed dentures).
  A 3rd appointment will be used for wax try-in for the conventional pathway. For the digital pathway, participants will have a chance to appraise their smile on a computer screen (virtual try-in, done remotely) and request modifications.
  Denture bases will be manufactured with conventional heat-polymerized resins, and participants will return for a 4th appointment for delivery, including chairside pick-up of attachments (GC Reline resin). Two short-term adjustments will be scheduled 24-72 h and 7 days after delivery, and then weekly until the dentures are comfortable.
  Interventions: Other: mandibular implant-overdenture

INTERVENTIONS:
Other: mandibular implant-overdenture — Mandibular overdentures fabricated over two implants will be delivered to the patients. In the first group, the 3D printed overdentures will be given for 3 months, followed by 3-month wear of traditional overdentures. The second group will wear traditional overdenture first followed by 3 months of 3D printed overdenture.

SUMMARY:
CAD/CAM (computer-aided design and computer-aided manufacturing) can be a game-changer for better access to care by edentulous patients. Digital overdentures offer potential for more satisfied patients due to better fit and can be provided faster/with lower costs. Providing digital overdentures has potential to enhance access to oral healthcare by the elderly, given the expected benefits (better quality, simpler, faster and more affordable than those obtained traditionally). However, evidence from randomized trials is crucial to verify the relevance of those benefits, especially from the patient perspective, and to confirm those benefits. This trial also serves as an opportunity to improve CAD software and materials, since it will identify technical challenges specific to the provision of digital overdentures.

This randomized cross-over trial aims to reveal whether implant-retained mandibular overdentures (IMO) produced by CAD and 3D printing are more satisfactory to edentulous seniors than those fabricated using traditional methods.

The investigators will recruit 26 edentulous participants (any sex/gender) amongst previous patients at McGill University, based on the following eligibility criteria: complete edentulism, elderly (age ≥60 years, according to the WHO), need for new maxillary and mandibular complete dentures, ability to complete questionnaires, and previous treatment with two implants in the anterior mandible. Each participant will receive two pairs of dentures, as per the McGill Consensus on Implant Overdentures (i.e., a mandibular overdenture opposed by a maxillary complete denture: (i) one by digital rendering of the mouth, virtual prosthetic design and 3D printing; (ii) a control pair, by traditional clinical and laboratory methods. Each pair will be worn for 3 months according to a random sequence (total follow-up: 6 months after the delivery of the first pair of dentures). Both overdentures will be retained by 2 Novaloc abutments and medium retention matrices.

Outcomes will include patient satisfaction ratings and oral health-related quality of life. The investigators will evaluate other patient-reported outcomes, as well as clinician-assessed quality and cost. Outcome assessment will occur at baseline, then at three months after participants have worn each pair of dentures. Following the cross-over, participants will keep their preferred denture pair and return after 12 months to evaluate maintenance requirements, including stained and broken dentures.

ELIGIBILITY:
Inclusion criteria:

* elderly according to the age cut-off purported by the World Health Organization (age >=60 years) and living independently;
* completely edentulous;
* no tooth extraction within the past 12 mo;
* two Straumann tissue level RN implants symmetrically distributed in the anterior mandible for 3 or + mo before the trial interventions;
* desire to receive both upper denture and lower IMO with new stud attachments;
* good understanding of spoken and written English or French;
* Ability to provide written informed consent.

Exclusion criteria:

* severe systemic disease or needing frequent hospitalization (i.e. American Society of Anesthesiologists Physical Status class >II);
* evidence of cognitive or motor impairment;
* acute or chronic symptoms of parafunctional or temporomandibular disorders;
* intraoral pathologies, either acute, progressive, potentially malignant or capable to hamper denture fit;
* signs of endosseous lesions or residual dental structures in panoramic radiographs;
* signs of implant failure, including clinical mobility, peri-implant radiolucency, unacceptable bone loss (0.2mm/year after 1st year, or <2mm any time) and persistent signs/symptoms (pain, neuropathy, infection or exudate).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Patient general satisfaction with full dentures | Baseline and after 3 months of wearing each denture
  The investigators will use the McGill Denture Satisfaction Questionnaire (MDSQ) to measure overall satisfaction (primary outcome), and satisfaction with specific aspects of the dentures - ability to chew, comfort, stability, aesthetics, ability to speak, and ability to clean

SECONDARY OUTCOMES:
Oral health related quality of life (OHQoL) | Baseline and after 3 months of wearing each denture
  This will be assessed by the OHIP-EDENT questionnaire
Clinical denture quality | Baseline and after 3 months of wearing each denture
  This trial will use the Functional Assessment of Dentures (FAD) instrument to assess denture quality from clinicians' perspective
Cost | through study completion, an average of 1 year
  The investigators will gather data on both the direct and indirect costs of each denture fabrication method
Qualitative report of adverse effects and maintenance needs. e.g. broken or stained dentures | through study completion, an average of 1 year
  The investigators will record all adverse events during the RCT at each post-delivery appointment and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University, Faculty of Dentistry, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
IDP will be shared according to the regulations set by McGill University, by the McGill Dataverse collection (available at: https://www.mcgill.ca/library/services/data-services/sharing )
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Scheduled at the moment of study completion (Anticipated: September 1, 2025)
URL: https://www.mcgill.ca/library/services/data-services/sharing

REFERENCES:
- [Derived] Jafarpour D, El-Amier N, Feine J, Bedos C, Abi-Nader S, Esfandiari S, Shuster T, Zimmermann E, de Souza R. 3D printing vs traditional workflow for the fabrication of mandibular implant overdentures: study protocol for a mixed-methods cross-over RCT. Trials. 2024 Apr 16;25(1):267. doi: 10.1186/s13063-024-08097-7. PMID 38627819